CLINICAL TRIAL: NCT00136318
Title: Efficacy and Tolerability of Escitalopram for the Prevention of Pegylated Interferon Alfa Associated Depression in Patients With Chronic Hepatitis C Infection: a Randomized Controlled Trial.
Brief Title: Escitalopram for the Prevention of PEGASYS-associated Depression in Hepatitis C Virus-infected Patients
Acronym: CIPPAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, M. Schaefer, MD, Martin Schaefer, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ML18075
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Depression
Keywords: Pegasys-Induced depression
MeSH Terms: conditions — Depression | interventions — Escitalopram; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator): After the preobservation period,patients received escitalopram, 10 mg per day. During treatment period, all patients began receiving antiviral therapy with PEG-interferon plus ribavirin with continuous concomitant administration of escitalopram.
  Interventions: Drug: Escitalopram; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Placebo (Placebo Comparator): After the preobservation period, patients received placebo. After 2 weeks of antidepressant pretreatment, all patients began receiving antiviral therapy with PEG-interferon plus ribavirin with continuous concomitant administration of placebo.
  Interventions: Drug: Placebo; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Escitalopram
  Arms: Escitalopram
Drug: Placebo
  Arms: Placebo
Drug: Peginterferon alfa-2a — Patients with HCV genotype 1 or 4 received treatment for 48 weeks with PEGinterferon-alfa2a, 180 mcg weekly. Patients with genotype 2 or 3 received PEGinterferon-alfa2a, 180 mcg weekly.
  Other Names: PEG-IFN alfa-2a; Pegasys
Drug: Ribavirin — Patients with HCV genotype 1 or 4 received treatment for 48 weeks with ribavirin, 1000 mg per day (body weight 75 kg) or 1200 mg per day (body weight, 75 kg). Patients with HCV genotype 2 or 3 received ribavirin, 800 mg per day for 24 weeks.

SUMMARY:
Primary end points

* incidence of depression defined as a Montgomery Asberg Depression Scale Score (MADRS) of 13 or higher during antiviral therapy (up to 48 weeks, depending on genotype)
* effect of an antidepressive pre-treatment over two weeks and a continuously concomitant treatment with Escitalopram (S-citalopram) on frequency and severity of depression in patients with chronic hepatitis C (HCV) treated with Peg-interferon alfa-2a (PEGASYS) and ribavirin, measured by the Montgomery Asberg Depression Scale

Secondary end points

* time to depression defined as a MADRS score of 13 or higher
* incidence of major depression defined by Diagnostic and Statistical Manual IV (DSM-IV) criteria
* severe depression according to MADRS scale (score 25 or higher)
* Health related quality of life (HRQOL) measured by the Short Form 36 (SF-36)
* sustained virologic response
* tolerability
* safety
* changes/group differences in other psychiatric depression scales (Hamilton Depression Rating Scale, Beck Depression Inventory)

Other investigations:

* cognitive function, anxiety (word fluency test, trail making test part A and B, othe scales)
* Predictive parameters for patients especially gaining from an antidepressive therapy (e.g. age, gender, weight, height, alanine aminotransferase (ALAT) quotient defined as median ALAT values before treatment divided by the upper standard value, HCV-RNA serum concentration level of fibrosis in liver histology, baseline values of the different psychometric scales)
* alanine aminotransferase (ALAT), aspartate transaminase (ASAT), thyrotrophin (TSH)
* biomarkers (genetic parameters, cytokines,...)

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection defined as positive anti-HCV antibodies and serum HCV-RNA >1000 IU/ml, naive to antiviral treatment
* age >18 years

Exclusion Criteria:

* Antidepressive treatment within the last 3 years
* Psychiatric diseases including major depressive disorders in past medical history
* Active substance abuse during the last 12 months
* Pregnancy, lactation, wish to become pregnant
* Hepatitis B (HBV)/HIV-coinfection
* Decompensated liver disease, hepatocellular carcinoma, history of bleeding esophageal varices
* Neutropenia (<1500/ul), thrombocytopenia (<70/nl), anemia (<12g/dl in females, <13g/dl in males)
* History of autoimmune disease
* History of organ transplantation, concomitant liver disease, severe cardiopulmonary disease, hemolytic anemia, malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2004-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berg, Prof. Dr., Study Chair — Charité; Martin Schaefer, Prof. Dr., Study Chair — Charite University, Berlin, Germany
Locations (1):
- Department of Gastroenterolgy and Rheumatology, Sektion Hepatology, Leipzig, Germany

REFERENCES:
- [Derived] Sarkar S, Sarkar R, Berg T, Schaefer M. Sadness and mild cognitive impairment as predictors for interferon-alpha-induced depression in patients with hepatitis C. Br J Psychiatry. 2015 Jan;206(1):45-51. doi: 10.1192/bjp.bp.113.141770. Epub 2014 Oct 30. PMID 25359924
- [Derived] Schaefer M, Sarkar R, Knop V, Effenberger S, Friebe A, Heinze L, Spengler U, Schlaepfer T, Reimer J, Buggisch P, Ockenga J, Link R, Rentrop M, Weidenbach H, Fromm G, Lieb K, Baumert TF, Heinz A, Discher T, Neumann K, Zeuzem S, Berg T. Escitalopram for the prevention of peginterferon-alpha2a-associated depression in hepatitis C virus-infected patients without previous psychiatric disease: a randomized trial. Ann Intern Med. 2012 Jul 17;157(2):94-103. doi: 10.7326/0003-4819-157-2-201207170-00006. PMID 22801672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 208 of the 300 patients screened were enrolled between August 2004 and September 2008 in different centers in the pre-observation period. Overall 181 patients started the treatment period by taking escitalopram or placebo.
Pre-assignment Details: A total of 208 of the 300 patients screened were enrolled between August 2004 and September 2008. 92 patients did not meet the inclusion criteria, had exclusion criteria or did not want to participate in the trial.27 patients stopped the trial during the preobservation period before the trial started by taking antidepressant or placebo therapy.
Groups:
- Escitalopram: After the preobservation period,patients received escitalopram, 10 mg per day. During treatment period, all patients began receiving antiviral therapy with PEG-interferon plus ribavirin with continuous concomitant administration of escitalopram.
  Peginterferon alfa-2a :
  Escitalopram :
  Ribavirin :
- Placebo: After the preobservation period, patients received placebo. After 2 weeks of antidepressant pretreatment, all patients began receiving antiviral therapy with PEG-interferon plus ribavirin with continuous concomitant administration of placebo.
  Peginterferon alfa-2a :
  Placebo :
  Ribavirin :
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 90 (Took first dose of study medication) | 91 (Took first dose of study medication)
Completed | 83 (reached end-point of antiviral treatment) | 84
Not Completed | 7 | 7
Not completed — Adverse Event | 5 | 5
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 84 | 168
  >=65 years | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11) | 48.5 (11) | 47.4 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 85
  Male | 48 | 48 | 96
Region of Enrollment [Number; unit: participants]
  Germany | 90 | 91 | 181

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Scale (MADRS) With a Score of 13 or Higher
Description: Clinically relevant depression (MADRS score of 13 or higher) during antiviral treatment presented as "percentage of participants" with "MADRS scores > 13" (entire time period: from starting study medication until end of antiviral treatment = 48 weeks in patients with genotype 1 or 4 and 24 weeks for patients with genotype 2 or 3)
Time Frame: 50 weeks for genotypes 1 or 4 and 26 weeks for patients with genotype 2 or 3
Population: The final analysis included only patients who received at least one of escitalopram or placebo. Between group differences for the primary outcome parameters were calculated with a chi-square test. For the primary end point (MADRS score of 13 or higher), we treated missing MADRS assessments by multiple imputation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Escitalopram: After the preobservation period, patients received escitalopram, 10 mg per day. During treatment period, all patients began receiving antiviral therapy with PEG-interferon plus ribavirin with continuous concomitant administration of escitalopram.
  Peginterferon alfa-2a :
  Escitalopram :
  Ribavirin :
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 90 | 91
percentage of participants | 32 [21 to 43] | 59 [48 to 69]

2. Secondary Outcome: Proportion of Patients Without Depression (Defined as a MADRS Score of 13 or Higher)
Description: Number of patients who did not develop at any time of antiviral treatment (up to 48 weeks) a MADRS score of 13 or more as a sign of clinically relevant depression
Time Frame: Patients free of depression during 24 or 48 weeks of antiviral therapy
Population: Number of patients per group who did not develop any depressive episode during 48 weeks of antiviral therapy.
Measure: Number; unit: participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 90 | 91
participants | 60 | 40

3. Secondary Outcome: Incidence of Major Depression Defined by Diagnostic and Statistical Manual IV (DSM-IV) Criteria
Time Frame: major depression during 24 or 48 weeks of antiviral therapy
Population: The final analysis included only patients who received at least 1 dose of escitalopram or placebo. Between-group differences for the secondary outcome parameters were calculated with a chi-square test.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 90 | 91
percentage of participants | 8 [4 to 15] | 17 [12 to 28]

4. Secondary Outcome: Severe Depression Defined as a MADRS Score of 25 or Higher
Time Frame: severe depression during 24 or 48 weeks of antiviral therapy
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 90 | 91
percentage of participants | 1 [0.3 to 6] | 12 [7 to 21]

5. Secondary Outcome: Health Related Quality of Life (HRQOL) Measured by the Short Form 36 (SF-36)
Time Frame: assessed 2,4,12,24 and 48 weeks of antiviral treatment
Reporting Status: Not Posted

6. Secondary Outcome: Sustained Virologic Response
Description: (negative Polymerase Chain Reaction (PCR) 6 months after the end of antiviral treatment)
Time Frame: assessed 24 weeks after end of antiviral treatment
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 90 | 91
percentage of participants | 56 [46 to 66] | 46 [37 to 57]

7. Secondary Outcome: Tolerability
Time Frame: assessed 2,4,12,24 and for genotype 1 and 4, 48 weeks of antiviral treatment
Reporting Status: Not Posted

8. Secondary Outcome: Safety
Time Frame: assessed 2,4,12,24 and for genotype 1 and 4, 48 weeks of antiviral treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 5/90 | 5/91
Other Adverse Events (participants affected / at risk) | 67/90 | 78/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=90) | Placebo (N=91)
drug abuse (Psychiatric disorders) | 1 | 0
self-harming behavior (Psychiatric disorders) | 1 | 0
renal failure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
cerebral tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
jaundice (General disorders) | 1 | 0
retinopathy (Eye disorders) | 0 | 1
glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
severe depression (Psychiatric disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=90) | Placebo (N=91)
Fatigue (General disorders) | 44 | 55
Dizziness (General disorders) | 13 | 23
Anemia (General disorders) | 16 | 20

LIMITATIONS AND CAVEATS:
Random assignment of patients before the preobservation period followed by patient withdrawal from the trial independent of antidepressant treatment weakens the strength of the randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No